CLINICAL TRIAL: NCT03009929
Title: International Multicentre Cohort Study for the External Validation of ClassIntra® - Classification of Intraoperative Adverse Events
Brief Title: Validation Study of ClassIntra®
Acronym: ClassIntra®
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00469
Record Dates: First submitted 2016-12-19; First posted 2017-01-04 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Patient Safety; Intraoperative Complications; Postoperative Complications; Risk Management
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Observational study — No intervention, observational only
  Other Names: No intervention, observational only

SUMMARY:
Whereas there are several validated systems for reporting postoperative complications, there are only a few and not prospectively validated systems for reporting intraoperative complications. The investigators developed a definition and CLASSification for Intraoperative Complications CLASSIC within a Delphi study involving international interdisciplinary experts. As both surgery and anaesthesia may be involved in complications in the perioperative period, all patient-related intraoperative complications occurring between skin incision and closure are considered in this reporting system. CLASSIC was updated to ClassIntra® v1·0, by encompassing five severity grades to align with the validated Clavien-Dindo Classification for grading postoperative complications.

The aim of this international multicentre observational cohort study is to assess the validity and practicability of this newly derived and updated classification system ClassIntra® in patient undergoing an in-hospital surgical procedure. Providing an easy applicable and internationally validated classification system is a contribution to improve quality of health care and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* All in-hospital patients (consecutive or random sample) undergoing surgery in the operating room with anaesthesia involvement

Exclusion Criteria:

* Outpatients (patients undergoing one-day-surgery) (with and without anaesthesia-involvement)
* Procedures without anaesthesia-involvement (in- or out-patient)
* ASA risk classification (ASA) VI patients (brain-death organ-donor)

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All in-hospital patients (consecutive or random sample) undergoing surgery in the operating room with anaesthesia involvement
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
intraoperative complications according to ClassIntra® | during surgery (intraoperatively)
  All intraoperative complications are recorded and classified according to their severity

SECONDARY OUTCOMES:
in-hospital postoperative complications | From after surgery up to hospital discharge, timeframe up to 30 days
  All postoperative complications observed during the hospital stay are recorded and classified according to their severity
Duration of surgery | From start to the end of the surgical procedure
  Time from start to end of the surgical procedure
Complexity of main surgical procedure | Baseline
  Complexity according to British United Provident Association (BUPA) classification
in-hospital mortality | From after surgery up to hospital discharge, timeframe up to 30 days
30-day mortality | 30 days postoperatively
Agreement in assessment of intraoperative complications between several raters using fictitious clinical case-scenarios using a questionnaire among physicians | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Salome Dell-Kuster, MD MSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (18):
- Carolinas Healthcare System, Charlotte, North Carolina, United States
- Northern Sydney Colorectal Clinic, Sydney, Australia
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Barmherzige Brüder Krankenhaus, Vienna
- Medical School, Aristotle University Thessaloniki, Thessaloniki, Greece
- Trinity College Dublin at Tallaght, Dublin, Ireland
- National Cancer Institute, Naples, Italy
- Radboud University Medical Centre, Nijmegen, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Hospital Valle de Hebron, Barcelona, Spain
- Switzerland (6):
  - University Hopsital Basel, Basel, Canton of Basel-City
  - University Childrens Hospital Basel, Basel
  - Kantonsspital Graubünden, Chur
  - University Hospital Lausanne, Lausanne
  - Bürgerspital Solothurn, Solothurn
  - Schulthess Clinique Zurich, Zurich
- Ankara University Medical School, Ankara, Turkey (Türkiye)
- Guy's and St. Thomas Hospital, London, United Kingdom

REFERENCES:
- [Derived] Gawria L, Rosenthal R, van Goor H, Dell-Kuster S; ClassIntra Study Group. Classification of intraoperative adverse events in visceral surgery. Surgery. 2022 Jun;171(6):1570-1579. doi: 10.1016/j.surg.2021.12.011. Epub 2022 Feb 15. PMID 35177252
- [Derived] Dell-Kuster S, Gomes NV, Gawria L, Aghlmandi S, Aduse-Poku M, Bissett I, Blanc C, Brandt C, Ten Broek RB, Bruppacher HR, Clancy C, Delrio P, Espin E, Galanos-Demiris K, Gecim IE, Ghaffari S, Gie O, Goebel B, Hahnloser D, Herbst F, Ioannidis O, Joller S, Kang S, Martin R, Mayr J, Meier S, Murugesan J, Nally D, Ozcelik M, Pace U, Passeri M, Rabanser S, Ranter B, Rega D, Ridgway PF, Rosman C, Schmid R, Schumacher P, Solis-Pena A, Villarino L, Vrochides D, Engel A, O'Grady G, Loveday B, Steiner LA, Van Goor H, Bucher HC, Clavien PA, Kirchhoff P, Rosenthal R. Prospective validation of classification of intraoperative adverse events (ClassIntra): international, multicentre cohort study. BMJ. 2020 Aug 25;370:m2917. doi: 10.1136/bmj.m2917. PMID 32843333